CLINICAL TRIAL: NCT06981637
Title: Maintenance Pegylated Liposomal Doxorubicin (PLD) Versus Active Surveillance for Advanced Soft Tissue Sarcoma Patients Who Had Controlled Disease After Standard Anthracycline-based Treatment (MELODY)
Brief Title: Pegylated Liposomal Doxorubicin (PLD) Versus Active Surveillance for Advanced Soft Tissue Sarcoma Patients Who Had Controlled Disease After Standard Anthracycline-based Treatment (MELODY)
Acronym: MELODY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Chang Gung Memorial Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); National Cheng-Kung University Hospital (Other); Tri-Service General Hospital (Other); China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T1725
Record Dates: First submitted 2025-05-05; First posted 2025-05-21 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Advanced Soft Tissue Sarcoma
Keywords: advanced soft tissue sarcoma; pegylated liposomal doxorubicin; open label randomized
MeSH Terms: interventions — liposomal doxorubicin

STUDY DESIGN:
Intervention Model Description: An investigator-initiated,A multinational open label randomized (2:1 experimental vs control) phase II study.
  Stratified randomization factor：
  1. The response after first-line anthracycline-based treatment (CR/PR vs SD)
  2. The study country.
  Patients will be randomized 2:1 using the method of minimization accounting for the stratification factors above.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pegylated liposomal doxorubicin (Experimental): Patients in experimental arm will receive pegylated liposomal doxorubicin (PLD) 40mg/m2 every 4 weeks. Maintenance PLD could be administered up to a total of 12 cycles.
  Interventions: Drug: Pegylated liposomal doxorubicin
- Active surveillance (No Intervention): Patients in control arm will receive active surveillance without treatment (treatment holiday). In control arm, crossover is not permitted after disease progression

INTERVENTIONS:
Drug: Pegylated liposomal doxorubicin — pegylated liposomal doxorubicin 40mg / m2 every 4 weeks for a maximum of 12 cycles.
  Other Names: Lipodox
  Arms: Pegylated liposomal doxorubicin

SUMMARY:
Maintenance Pegylated Liposomal Doxorubicin (PLD) Versus Active Surveillance for Advanced Soft Tissue Sarcoma Patients Who Had Controlled Disease After Standard Anthracycline-based Treatment (MELODY)

DETAILED DESCRIPTION:
Patients enrolled will be randomized to either experimental arm or control arm. Patients in experimental arm will receive pegylated liposomal doxorubicin (PLD) 40mg/m2 every 4 weeks. Maintenance PLD could be administered up to a total of 12 cycles. Patients in control arm will receive active surveillance without treatment (treatment holiday).

ELIGIBILITY:
Inclusion Criteria:

1. A histologically confirmed advanced soft tissue sarcoma. Note that subtypes typically do not use chemotherapy as standard treatment are not allowed, such as alveolar soft part sarcoma, solitary fibrous tumor, extraskeletal myxoid chondrosarcoma, clear cell sarcoma)
2. Patients received first-line anthracycline-based treatment for a minimum of 4 cycles and a maximum of 8 cycles.
3. The best response after first-line anthracycline-based treatment must be either a complete response, partial response, or stable disease as defined by RECIST 1.1.

   The best response should be attributed solely to systemic treatment and not to local therapy. All the patients must have at least one measurable tumor based on RECIST 1.1 before initiating first-line anthracycline-based treatment.
4. Patients must be randomized within 8 weeks of their last dose of anthracycline-based treatment
5. Patients have a life expectancy ≥ 3 months
6. Patients older than 18 years old.
7. ECOG performance status of 0 to 1.
8. Patients must have adequate organ function and marrow reserve measured within 7 days prior to randomization as defined below:

   1. Hemoglobin ≥ 9.0 g/dL;
   2. Absolute neutrophil count ≥ 1,500/mm3;
   3. Platelets ≥ 100,000/mm3;
   4. Total bilirubin ≤ 1.5 x upper normal limit;
   5. AST(SGOT)/ALT(SGPT) ≤ 2.5 x upper normal limit; for patients with liver metastases AST(SGOT)/ALT(SGPT) ≤ 5 x upper normal limit is allowed;
   6. Serum creatinine ≤ 1.5mg/dL or creatinine clearance ≥50ml/min;
   7. All women of childbearing potential must have a negative pregnancy test obtained within 72 hours before starting therapy.
9. For male participants: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm.
10. Patients with reproductive potential must use effective contraception (hormone orbarrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 months after the completion of therapy.
11. Patients must be able to comply with study procedures and sign informed consent.

Exclusion Criteria:

1. Known allergy history to PLD or other drugs of liposome-based formulation.
2. LVEF < 50% at screening as determined by UCG or MUGA.
3. Serious non-healing wound, ulcer, or bone fracture not related to underlying sarcoma.
4. Major surgical procedure, open biopsy, significant traumatic injury, or radiotherapy within 21 days prior to randomization.
5. Severe, uncontrolled medical conditions including severe liver disease, heart disease, uncontrolled diabetes or hypertension, or pulmonary disease.
6. Psychiatric illness or social situation that would preclude study compliance.
7. Women with pregnant or breast feeding (a urine pregnancy test must be performed on all female patients who are of childbearing potential before entering the study, and the result must be negative.
8. Another previous malignancy diagnosed within the past 3 years. Patients with carcinoma in situ and stage I malignancy under active surveillance (no medical treatment needed) are allowed for enrollment.
9. Active CNS metastasis defined by clinical symptoms, cerebral edema, steroid or anti- convulsant requirement, or progressive growth. Patients with a history of CNS metastasis or cord compression are allowed in the study if they have been treated and are clinically stable.
10. Patients with active hepatitis B. However, patients with controlled hepatitis B under anti-viral agent are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-12-31 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival from randomization | Up to approximately 2 years
  The Tumor response will be assessed according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1, see Appendix 2) every 8 weeks, and every 12 weeks 24 weeks after randomization.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 2 years
  Defined as the time from the date of randomization to the date of death from any cause, or censoring at the date of last known follow-up alive
Progression-free survival (PFS) | Up to approximately 2 years
  Progression-free survival (PFS) rate at 12 months. PFS is defined as the time from the date of randomization to the date of first documented evidence of progressive disease (including radiograph or clinical progressive disease), or death, whichever occurs first.
Time to next treatment (TTNT) | Up to approximately 2 years
  Defined as the time from the date of randomization to the date of commencing next treatment line. Patients who started other anti-cancer therapy (including radiotherapy and surgery) will be counted as an event for TTNT. Those who received radiotherapy or surgical resection after randomization but not based on clinical or radiological progression are considered as an event for TTNT.
Objective response rate (ORR) | Up to approximately 2 years
  Objective response rate (ORR) at maintenance PLD phase per RECIST 1.1 criteria
Frequency and severity of AE | Up to approximately 2 years
  AEs will be accessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).
Safety of interest: cardiac function as assessed by LVEF | Up to approximately 2 years
  Safety of interest: cardiac function as assessed by LVEF(either by cardiac US or MUGA)
Quality of Life Effects on patient-reported outcomes as assessed by EORTC QLQ C30 | Up to approximately 2 years
  The questionnaire comprises 5 functioning scales (physical, role, emotional, cognitive, and social functioning), 9 symptom scales (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties), and a global health status/QoL scale. The functioning and symptoms items are scored on a 4-point scale that range from "not at all" to "very much," and the global health status and QoL items are scored on a 7-point scale that ranges from "very poor" to "excellent.". There are 30 questions in total and the scores range from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Tsang-Wu Liu, MD, Study Director — Taiwan Cooperative Oncology Group, National Health Research Institutes; Tom Wei-Wu Chen, MD,PhD, Principal Investigator — National Taiwan University Hospital
Locations (7):
- Taiwan (7):
  - Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital,, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No